CLINICAL TRIAL: NCT05127421
Title: A Phase 2, Efficacy and Safety Study of Ruxolitinib Cream in Participants With Facial and/or Neck Atopic Dermatitis Involvement
Brief Title: Ruxolitinib Cream in Participants With Facial and/or Neck Atopic Dermatitis Involvement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-215
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; adolescent; adults; in-home; telemedicine
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: This is 2:1 assignment to rux and vehicle creams.
Who Masked: Participant, Investigator
Masking Description: 4 week double-blind treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Double-blind Period: vehicle cream or Ruxolitinib cream 1.5% BID (Experimental): Participants will be treated with ruxolitinib cream 1.5% or vehicle cream twice a day (BID) in a double-blind fashion.
  Interventions: Drug: Ruxolitinib cream; Drug: Vehicle
- Open Label Extension: Ruxolitiib cream 1.5% (Experimental): Patients will be treated with Ruxoltinib cream 1.5% twice per day (BID) during the open label extension period. Participants who complete the double-blind period will continue into this open-label extension period for an additional 4 weeks of treatment.
  Interventions: Drug: Ruxolitinib cream

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream 1.5% applied twice a day (BID)"
Drug: Vehicle — Vehicle cream applied twice a day (BID) to affected areas
  Arms: Double-blind Period: vehicle cream or Ruxolitinib cream 1.5% BID

SUMMARY:
This is a randomized, double blind, vehicle controlled Phase 2 study with a 4-week open label extension in adolescent and adult participants with atopic dermatitis and head and/or neck involvement. It is intended to compare the efficacy and safety of ruxolitinib cream 1.5% BID versus vehicle cream, then further evaluate ruxolitinib cream as maintenance during the open label extension period.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of AD for at least 6 months.
* Participants with an overall and a face and/or neck IGA score of 2 or 3 at screening and baseline.
* Participants with AD affecting the following at screening and baseline:

  1. ≥ 0.5% of the total BSA on the face and/or neck
  2. Up to a total of 20% BSA (face and/or neck plus other body areas)
* Willingness to avoid pregnancy or fathering children based on the criteria outlined in the protocol.
* Further inclusion criteria apply.

Exclusion Criteria:

* Participants who have an unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks prior to baseline.
* Participants with concurrent conditions and history of other diseases such as immunocompromised; chronic or acute infection requiring systemic treatments; active acute skin infection; other concomitant skin conditions that may interfere with the evaluation of AD or compromise participant safety; other types of eczema; chronic asthma requiring high dose of inhaled corticosteroids.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Previous treatment with systemic or topical JAK inhibitors (eg, ruxolitinib, tofacitinib, baricitinib, filgotinib, lestaurtinib, pacritinib).
* Participants who are pregnant (or who are considering pregnancy) or lactating.
* Laboratory values outside of the protocol -defined criteria
* Further exclusion criteria apply.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haq Nawaz, MD, Study Director — Incyte Corporation
Locations (1):
- Science37, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Chiesa Fuxench ZC, Lai Z, Kuo Y, Nawaz H, Cotliar J. Ruxolitinib cream monotherapy for facial and/or neck atopic dermatitis: results from a decentralized, randomized phase 2 clinical trial. J Dermatolog Treat. 2025 Dec;36(1):2480744. doi: 10.1080/09546634.2025.2480744. Epub 2025 Mar 25. PMID 40132224

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This decentralized clinical study was conducted through 1 virtual meta-site in the United States.
Groups:
- Double-Blind Period: Vehicle Cream BID: Participants applied matching vehicle cream BID for 4 weeks.
- Double-Blind Period: Ruxolitinib Cream 1.5% BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) for 4 weeks.
- Open-Label Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID: Participants who completed the Week 4 assessments with no safety concerns could continue into the 4-week Open-Label Period. Participants who applied vehicle cream BID during the Double-Blind Period applied ruxolitinib cream 1.5% BID for 4 weeks in the Open-Label Period.
- Open-Label Period: Ruxolitinib Cream 1.5% BID: Participants who completed the Week 4 assessments with no safety concerns could continue into the 4-week Open-Label Period. Participants who applied ruxolitinib cream 1.5% BID during the Double-Blind Period continued to apply ruxolitinib cream 1.5% BID for an additional 4 weeks in the Open-Label Period.
Period: 4-Week Double-Blind Period
Arm/Group | Double-Blind Period: Vehicle Cream BID | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Open-Label Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID | Open-Label Period: Ruxolitinib Cream 1.5% BID
Started | 23 | 54 | 0 | 0
Completed | 18 | 48 | 0 | 0
Not Completed | 5 | 6 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Not completed — Withdrawn by Sponsor | 0 | 4 | 0 | 0
Not completed — Withdrawn Due to E-diary Compliance | 0 | 1 | 0 | 0
Period: 4-Week Open-Label Period
Arm/Group | Double-Blind Period: Vehicle Cream BID | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Open-Label Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID | Open-Label Period: Ruxolitinib Cream 1.5% BID
Started | 0 | 0 | 17 | 47
Completed | 0 | 0 | 16 | 44
Not Completed | 0 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Withdrawn by Sponsor | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Period: Vehicle Cream BID | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Total
Number analyzed (Participants) | 23 | 54 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (13.44) | 37.9 (14.37) | 38.8 (14.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 46 | 62
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 22 | 49 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 11 | 20 | 31
  Black/African-American | 10 | 24 | 34
  Asian | 1 | 4 | 5
  American-Indian/Alaska Native | 0 | 1 | 1
  Black, Asian | 1 | 0 | 1
  Captured as "Hispanic" in the Database | 0 | 1 | 1
  Black and Phillipino | 0 | 1 | 1
  Mexican | 0 | 1 | 1
  Indian | 0 | 1 | 1
  Mexican and Spanish | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a ≥75% Improvement in the Eczema Area and Severity Index Score (EASI75) of the Head and Neck Region at Week 4
Description: The EASI scoring system examines 4 areas of the body (head/neck, trunk, upper limbs, and lower limbs) and weights them for participants of at least 8 years of age. Each of the 4 body regions is assessed separately for erythema (E), induration/papulation/edema (I), excoriations (Ex), and lichenification (l) on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72; the severity strata are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. Specifically for the head and neck region, the EASI score ranges from 0 to 7.2 An EASI75 responder was defined as a participant achieving a 75% or greater improvement from Baseline in the EASI score for the head and neck.
Time Frame: Baseline; Week 4
Population: Full Analysis Population: all participants enrolled in the study who had at least 1 application of study drug. Missing post-Baseline values were imputed as Non-Responders at Week 4. The 95% confidence interval for the difference was computed based on a large-sample normal approximation with continuity correction.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind Period: Vehicle Cream BID | Double-Blind Period: Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 23 | 54
percentage of participants | 17.4 [5.0 to 38.8] | 37.0 [24.3 to 51.3]
Statistical Analysis 1: Comparison: Double-Blind Period: Vehicle Cream BID vs Double-Blind Period: Ruxolitinib Cream 1.5% BID; Test type: Superiority; p = 0.091, Cochran-Mantel-Haenszel; stratified by the stratification factor (face and/or neck Investigator's Global Assessment [IGA] score of 2 or 3 at screening); Odds Ratio (OR) = 2.81, 95% CI 2-sided [0.83 to 9.47]
Statistical Analysis 2: Comparison: Double-Blind Period: Vehicle Cream BID vs Double-Blind Period: Ruxolitinib Cream 1.5% BID; Test type: Superiority; response rate difference = 19.5, 95% CI 2-sided [-0.5 to 39.6], Standard Error of Mean 10.23 — The 95% confidence interval was computed based on a large-sample normal approximation with continuity correction

2. Secondary Outcome: Percentage of Participants Who Achieve an EASI75 of the Head and Neck Region at Weeks 2 and 8
Description: as for outcome 1
Time Frame: Baseline; Weeks 2 and 8
Population: Full Analysis Population. Only participants with available data were analyzed. The 95% confidence interval for the difference was computed based on a large-sample normal approximation with continuity correction.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind Period: Vehicle Cream BID | Double-Blind Period: Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 18 | 48
percentage of participants
  Week 2 | 16.7 [3.6 to 41.4] | 14.6 [6.1 to 27.8]
  Week 8: number analyzed (Participants) | 17 | 45
  Week 8 | 35.3 [14.2 to 61.7] | 53.3 [37.9 to 68.3]

3. Secondary Outcome: Percentage of Participants Who Achieve an Overall EASI75 at Weeks 2, 4, and 8
Description: The EASI scoring system examines 4 areas of the body (head/neck, trunk, upper limbs, and lower limbs) and weights them for participants of at least 8 years of age. Each of the 4 body regions is assessed separately for erythema (E), induration/papulation/edema (I), excoriations (Ex), and lichenification (l) on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72; the severity strata are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. An EASI75 responder was defined as a participant achieving 75% or greater improvement from Baseline in EASI score.
Time Frame: Baseline; Weeks 2, 4, and 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind Period: Vehicle Cream BID | Double-Blind Period: Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 18 | 48
percentage of participants
  Week 2 | 5.6 [0.1 to 27.3] | 10.4 [3.5 to 22.7]
  Week 4: number analyzed (Participants) | 17 | 45
  Week 4 | 33.3 [13.3 to 59.0] | 29.2 [17.0 to 44.1]
  Week 8: number analyzed (Participants) | 17 | 45
  Week 8 | 35.3 [14.2 to 61.7] | 33.3 [20.0 to 49.0]

4. Secondary Outcome: Double-Blind Period: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any adverse event (AE) either reported for the first time or the worsening of a pre-existing event after the first application of the study drug. An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug.
Time Frame: up to approximately 4 weeks plus 30 days
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period: Vehicle Cream BID | Double-Blind Period: Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 23 | 54
Participants | 5 | 6

5. Secondary Outcome: Open-Label Period: Number of Participants With Any TEAE
Description: A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first application of the study drug. An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug.
Time Frame: from first dose date in Open-Label Period (start of Week 5) until last follow-up visit (up to approximately 4 weeks plus 30 days)
Population: Open-Label Evaluable Population: all participants who applied at least 1 dose of ruxolitinib cream during the Open-Label Period
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID | Open-Label Period: Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 17 | 47
Participants | 4 | 9

6. Secondary Outcome: Double-Blind Period: Number of Participants With Any Grade 3 or Higher TEAE
Description: A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first application of the study drug. An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. The severity of AEs was graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Grades 1 to 5). Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL). Grade 3: severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4: life-threatening consequences; urgent intervention indicated. Grade 5: death related to AE.
Time Frame: up to approximately 4 weeks plus 30 days
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period: Vehicle Cream BID | Double-Blind Period: Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 23 | 54
Participants | 0 | 1

7. Secondary Outcome: Open-Label Period: Number of Participants With Any Grade 3 or Higher TEAE
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Open-Label Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID | Open-Label Period: Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 17 | 47
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: from the time of Informed Consent Form signing until at least 30 days after the last application of study drug (up to Week 8 + 30 days)
Description: Treatment-emergent adverse events (TEAEs): AEs reported for the first time or the worsening of pre-existing events after the first application of study drug. For the Double-Blind Period, TEAEs are reported for members of the Full Analysis Population: all participants who had at least 1 application of study drug.. For the Open-Label Period, TEAEs are reported for the Open-Label Evaluable Population: all participants who applied at least 1 dose of ruxolitinib cream during the Open-Label Period.
Groups:
- Vehicle Cream BID: Participants applied matching vehicle cream twice a day (BID) for 4 weeks in the Double-Blind Period.
- Ruxolitinib Cream 1.5% BID: Participants applied ruxolitinib cream during the Double-Blind Period and the Open-Label Period. Participants who completed the Week 4 assessments with no safety concerns could continue into the 4-week Treatment-Extension Period. Participants who applied ruxolitinib cream 1.5% BID during the Double-Blind Period continued to apply ruxolitinib cream 1.5% BID for an additional 4 weeks in the Open-Label Period. Participants who applied vehicle cream BID during the Double-Blind Period applied ruxolitinib cream 1.5% BID for 4 weeks in the Open-Label Period.
Arm/Group | Vehicle Cream BID | Ruxolitinib Cream 1.5% BID
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/71
Other Adverse Events (participants affected / at risk) | 2/23 | 1/71
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=23) | Ruxolitinib Cream 1.5% BID (N=71)
Application site reaction (General disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT05127421/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT05127421/SAP_001.pdf